CLINICAL TRIAL: NCT05203133
Title: Investigating the Combined Effect of Acute Energy Deficit and Aerobic Exercise Training on Muscle Quality in Healthy Adult Males
Brief Title: Effects of Acute Energy Deficit and Aerobic Exercise on Muscle Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 21LJMUSPONSOR052
Record Dates: First submitted 2021-09-28; First posted 2022-01-24 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Energy Supply; Deficiency; Energy Balance; Energy Availability
Keywords: Dynamic proteomic profile; Skeletal muscle; Intra-muscular lipid profiles; Skeletal muscle glycogen; Glucose; Insulin; Leptin; Ghrelin; Testosterone; Adiponectin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants will complete a 5-day free-living baseline assessment period (days -5 to -1) and two consecutive 5-day periods (days 1 - 10, with a final assessment on the morning of day 11) of controlled exercise to increase oxidative capacity (3 days of aerobic exercise per period, 15 kcal/kg FFM/day energy expenditure cycling) and energy intake.
  This will achieve states of energy balance (EB; energy availability - EA - 45 kcal/kg of fat free mass (FFM)/day), required for weight maintenance (days 1 - 5), followed by energy deficit (ED; EA 10 kcal/kg FFM/day), required for weight loss on days 6 - 10.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline Assessment (Days -5 to -1) (Experimental): Participants will complete a a 5-day baseline assessment in which habitual energy intake (remote food photography method) and exercise energy expenditure will be monitored.
  Interventions: Dietary Supplement: Baseline Assessment
- Energy Balance (Days 1 to 5) (Experimental): Participants will be provided with all food intake for five days, to provide an energy intake of 54 kcal/kg FFM/day. On days 1, 3 and 5, participants will complete aerobic (cycling) exercise at ~60% VO2peak to expend15 kcal/kg FFM. This will achieve a state of energy balance (energy availability = 45 kcal/kg of FFM/day, required for weight maintenance.
  Interventions: Dietary Supplement: Energy Balance
- Energy Deficit (Days 6-11) (Experimental): Participants will be provided with all food intake for five days, to provide an energy intake of 19 kcal/kg FFM/day. On days 6, 8 and 10, participants will complete aerobic (cycling) exercise at ~60% VO2peak to expend15 kcal/kg FFM. This will achieve a state of energy deficit (energy availability = 10 kcal/kg of FFM/day) resulting in ~2.5 kg of weight-loss.
  Interventions: Dietary Supplement: Energy Deficit

INTERVENTIONS:
Dietary Supplement: Energy Balance — Energy balance phase to elicit weight-maintenance
  Arms: Energy Balance (Days 1 to 5)
Dietary Supplement: Energy Deficit — Energy deficit phase to elicit weight-loss
  Arms: Energy Deficit (Days 6-11)
Dietary Supplement: Baseline Assessment — Free-living assessment of energy status
  Arms: Baseline Assessment (Days -5 to -1)

SUMMARY:
10 healthy, male, participants will complete a a 5-day baseline assessment (days -5 to -1) and two consecutive 5-day periods of controlled exercise to increase oxidative capacity (3 days of aerobic exercise per period, 15 kcal/kg FFM/day energy expenditure cycling) and energy intake (15 days in total, with a testing session on morning 16). This will achieve states of energy balance (EB; energy availability - EA - 45 kcal/kg of fat free mass (FFM)/day), required for weight maintenance (days 1 - 5), followed by energy deficit (ED; EA 10 kcal/kg FFM/day), required for weight loss on days 6 - 10.

Over the data-collection period, participants will consume deuterium (D2O) tracer to facilitate dynamic proteomic profiling to assess the impact of the intervention on muscle quality (primary outcome measure). Muscle biopsies will therefore be collected on days -5, 1, 6 & 11, alongside daily saliva samples, and venous blood collection on days -5, 1, 3, 5, 6, 8, 10 & 11. These samples will be used to assess further, secondary, outcome measures including alterations in intra-muscular lipid profiles (lipid droplet content, morphology and lipid-droplet associated proteins in different subcellular compartments [intermyofibrillar vs subsarcolemmal]), alterations in blood metabolites and hormones and skeletal muscle glycogen concentrations. Changes in body mass, body composition and RMR will also be assessed.

DETAILED DESCRIPTION:
Justification for the research:

Weight-loss strategies that use energy restriction alone can lead to impaired muscle mass, which can also further impair health of individuals with metabolic conditions, such as type 2 diabetics. Skeletal muscle mass and function are key to maintaining a healthy metabolism and quality of life throughout the lifespan. The combination of exercise and calorie restriction is a powerful intervention for reducing body weight and improving the metabolism and health status of healthy, overweight and obese individuals. The investigators have previously shown that skeletal muscle protein synthesis is reduced with energy restriction and that resistance-type exercise can reverse this negative effect. Aerobic-type exercise also has the capacity to stimulate muscle protein synthesis and improve the quality of muscle by increasing mitochondrial protein synthesis. Nonetheless, how energy deficit overlayed on top of aerobic exercise modulates skeletal muscle quality is not well characterised. Furthermore, existing studies have looked only into mixed (unspecific) protein synthesis of different intracellular compartments without providing details on how protein synthesis for specific proteins is regulated.

This project will provide novel data to unravel the mechanisms behind the positive effect of energy restriction and concomitant aerobic exercise on skeletal muscle quality.

Aerobic exercise alone is a well-established intervention to increase mitochondrial capacity and skeletal muscle function, but the effect on skeletal muscle of overlaying energy restriction while performing aerobic exercise is not well characterised. Recent findings in Rhesus monkeys, whose physiology responds in a very similar way to that of humans, has shown that life-long caloric restriction has a profound positive effect on skeletal muscle. These findings show that caloric restriction not only maintains contractile content of muscle, but also rescues the age-related decline of skeletal muscle mitochondrial content and capacity. However, physical activity in this study was not controlled and appeared to be higher in the caloric restriction group, representing an important confounding factor. Research in humans addressing similar questions so far has been less clear. Pronounced weight loss through energy restriction alone (10% total body weight in ~7.5 wk) in obese women lead to a decrease in muscle mitochondrial content. In stark contrast, using a milder restriction of 25% of total energy alone or combined with exercise during 6 months in overweight individuals showed increased expression of genes encoding mitochondrial proteins in both groups. However, despite these promising findings suggesting that weight-loss combined with exercise will enhance skeletal muscle metabolism, there are currently no strong data to provide support on the use of concomitant energy restriction and aerobic exercise with in-depth analysis of its physiological and molecular effects in humans.

The proposed study herein will include a short period of tightly controlled exercise and dietary intake to show that energy deficit while performing aerobic exercise results in further benefits to muscle metabolic adaptation. The current project builds on from the investigator's previous and recent research findings to directly address this question. This research has shown that resistance exercise during 30% daily energy deficit rescues the decrease in mixed (unspecific) myofibrillar protein synthesis observed with energy deficit alone. Moreover, the investigator's research has shown that aerobic exercise up-regulates specific proteins in skeletal muscle mitochondria in rodents; that skeletal muscle lipid droplet profile is responsive to exercise and nutrition; that nutrition modulates the cellular response to aerobic exercise and, importantly; that aerobic exercise after short-term (~14 hours) energy deficit can up-regulate markers of mitochondrial biogenesis in skeletal muscle and improve metabolic control in humans.

Objectives & Hypothesis:

The primary research question associated with this study is: 'What is the combined effect of an energy deficit and aerobic exercise training on muscle quality (synthesis rates of individual, sarcoplasmic and mitochondrial proteins) and intramuscular lipid dynamics over a five-day period in healthy males?'

Further objectives:

1. Identify the mechanisms by which a short-term energy deficit (achieved through concomitant energy restriction and exercise) can regulate individual muscle protein turnover (synthesis, breakdown and abundance), intramuscular lipid dynamics, metabolites and muscle glycogen content during weight-loss.
2. Provide novel evidence for the capacity of a potato-based diet as an effective source of nutrients to promote positive skeletal muscle and metabolic adaptations during weight loss.

Study hypothesis:

Short-term energy restriction with concomitant aerobic exercise will increase the quality and quantity of skeletal muscle proteins related to mitochondrial capacity, improve skeletal muscle intracellular lipid droplet profile and modulate blood-borne markers of metabolic health compared to exercise without energy deficit.

Study Methods:

Participants will first undertake testing for characterisation (detailed below) followed by a 5-day baseline assessment (days -5 to -1) and two consecutive 5-day periods of controlled exercise to increase oxidative capacity (3 days of aerobic exercise per period, 15 kcal/kg FFM/day energy expenditure running) and energy intake (15 days in total, with a testing session on morning 16). This will achieve states of energy balance (EB; energy availability - EA - 45 kcal/kg of fat free mass (FFM)/day), required for weight maintenance (days 1 - 5), followed by energy deficit (ED; EA 10 kcal/kg FFM/day), required for weight loss on days 6 - 10. This experimental design, as well as energy intake and expenditure, replicates what the investigators have previously used to successfully determine other physiological effects of ED on skeletal muscle. Five days of EB and EA will allow for tight control of dietary intake and will be sufficient to detect changes in the main parameters being investigated.

Participant characterisation testing will be ~15 days prior to the start of baseline assessment to determine compliance with inclusion criteria, fitness levels (maximal oxygen consumption and lactate threshold [via finger-prick capillary samples]) and body composition. At baseline assessment a resting muscle a biopsy will be taken from the vastus lateralis (quadriceps), prior to ingestion of the tracer deuterium oxide (D2O) through the following 15 days to allow dynamic proteomic profiling of skeletal muscle. A total of 4 biopsies will be taken per participant, which is in line with the investigator's prior research. The baseline assessment is used for enrichment of D2O for dynamic proteomic profiling assay and ensuring regular physical activity of individuals matches requirements of the study. Throughout each 5-day experimental period, muscle biopsies (days -5, 1, 6 & 11), daily saliva samples (non-stimulated, collected at home) and regular venous blood samples (days -5, 1, 3, 5, 6, 8, 10 & 11) will be collected for the assessment of dynamic proteomic profiling, fibre-type specific lipid droplet profiling, skeletal muscle glycogen and D2O, and blood-borne hormones and metabolites related to weight loss. Resting Metabolic Rate (RMR; assessed via indirect calorimetry) and body composition assessment will be conducted using dual X-ray absorptiometry (DXA) scans on days -5, 1, 6 & 11 of the intervention. Bioelectrical impedance analysis (BIA) will also be used to assess body composition at each lab visit (days -5, 1, 3, 5, 6, 8, 10 & 11).

Dietary interventions and energy balance:

The diet will follow the reference daily intake of nutrients to provide ~60, 20 and 20% of energy from carbohydrates, fat and protein, respectively. In line with funding requirements, the percentage of total energy from potato-based sources will be >60% during EB and >65% during ED. Potatoes will be cooked in a range of different ways that do not add significant amount of energy such as boiled, microwaved, baked, etc.

Energy availability manipulation:

Energy availability (EA), which is defined as energy intake minus energy expenditure from exercise - normalised to fat free mass - is used as a key parameter to determine energy balance. The investigators are the first to have shown that values under 30 kcal/kg/FFM can modulate skeletal muscle responses, which is in line with other research on a range of metabolic responses to EA. Based on this recent research, which used 20 kcal/kg FFM/day for ~14 hs, the current intervention will induce a more pronounced energy deficit for longer. The average energy intake across the 5 days for an average 85 kg (70 kg FFM) participant will be 3780 kcal/day for EB and 1330 kcal/day ED. This will achieve an approximate cumulative energy deficit of 12250 kcal over the 5-day period resulting in approximately ~1.5 kg of body mass loss from net tissue, given that ~7450 kcal are necessary to lose 1 kg of net tissue. Water loss will account for an additional ~1 kg of the loss in body weight which will be a consequence of a decrease in endogenous carbohydrate (glycogen) stores, to which water binds, as well water fluctuation due to sodium changes. Skeletal muscle glycogen is also a regulator of the muscle qualitative aspects and will also be investigated.

Subjects. A normal population will allow the researchers to determine the physiological responses to this intervention. Ten young (18-40 years) healthy, regularly exercising men with a body fat percentage ~18-26%.

Quality:

The researcher's associated with this study and associated with the review of the study protocol are all members of staff (or a PhD Student) within the Liverpool John Moores University Research Institute for Sport & Exercise Sciences (RISES). In the 2014 RISES (LJMU) submitted 34.75 FTE (full time equivalent) to Unit of Assessment 26 (UoA26) and attained a GPA (Grade Point Average) of 3.57. Placed second on GPA in the UoA, RISES became the leading centre for Sport and Exercise Science Research Quality in the UK (4* - 61% of all activity world leading, 3* - 36% of all activity internationally excellent standard). RISES submitted the largest volume of 4* outputs (n=60) in the UoA, had 90% of the impact activity rated at 4* and had 100% of the environment rated as 4*. Importantly, out of 1,911 submissions in all 36 UoA's RISES came 11th in the entire UK for GPA achieved at REF2014 putting RISES (LJMU) amongst Oxford, UCL, LSE and Cambridge in the league tables for this metric.

ELIGIBILITY:
Inclusion Criteria:

* Gender/Sex - Male
* Age - 18 - 40
* % body fat - ~18 - 26 %
* Health - Healthy (as determined by pre-participation questionnaires)
* Training Status - Regularly Exercising/Aerobically trained (3-4 aerobic training sessions/week, 3-5 hrs/week) Non-smokers
* Weight-stable (within 2 kg) for the past 6-months

Exclusion Criteria:

* Gender/Sex - Female/Other
* Age - <18 - >40
* Health - Deemed unable to perform exercise (assessed via readiness to exercise questionnaire)
* Current smoker.
* Medical Condition - Those with any previous diagnosis of; Osteoporosis/low bone mineral density, cardio-vascular disease, Diabetes Mellitus, Cerebrovascular Disease, blood-related illness/disorder, Asthma or other respiratory illness/disorder, Liver Disease, Kidney Disease, gastrointestinal disease, Eating Disorder or Disordered Eating.
* Those currently taking prescription medication or unwell with a cold or virus at the time of participation.
* Those unwilling to adhere to the study's methodological requirements (including adhering to alterations in diet and training - inc. alcohol abstention) from the day prior to intervention onset (24 hrs pre-intervention) to completion of follow-up assessments (day-11).
* Those following a restrictive diet (e.g. vegetarians/vegans)
* Any individuals with a food allergy/intolerance
* Training status - Does not train aerobically 3 + times/week (over past 6 months on average)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Alterations to skeletal muscle proteome | Days -5, 1, 6 & 11
  Quantification of changes in skeletal muscle quality via dynamic proteomic profiling following short-term energy balance and energy deficit.

SECONDARY OUTCOMES:
Intra-muscular lipid profile: lipid droplet content | Days -5, 1, 6 & 11
  Assessment of alterations in intra-muscular lipid droplet content
Intra-muscular lipid profile: lipid droplet morphology | Days -5, 1, 6 & 11
  Assessment of alterations in intra-muscular lipid morphology
Intra-muscular lipid profile: lipid droplet associated proteins | Days -5, 1, 6 & 11
  Assessment of alterations in intra-muscular lipid-droplet associated proteins
Blood metabolites/hormones: Glucose concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Blood metabolites/hormones: Insulin concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Blood metabolites/hormones: Leptin concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Blood metabolites/hormones: Ghrelin concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Blood metabolites/hormones: Lactate concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Blood metabolites/hormones: Testosterone concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Blood metabolites/hormones: Adiponectin concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Blood metabolites/hormones: Triiodothyronine concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Blood bone turnover markers: Beta-CTX concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Blood bone turnover markers: P1NP concentrations | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in blood metabolites and hormones following short-term energy balance and energy deficit.
Skeletal Muscle Glycogen Concentrations | Days -5, 1, 6 & 11
  Assessment of alterations in skeletal muscle glycogen concentrations following short-term energy balance and energy deficit.
Changes in body composition: Body Mass (kg) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Body Mass Index [BMI] (kg/m^2) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Fat Mass (kg) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Body Fat Percentage (%) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Fat Free Mass (kg) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Skeletal Muscle Mass (kg) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Total Body Water (l) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Total Body Water (%) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Extracellular Water (l) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Extracellular Water (%) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Extracellular Water/Total Body Water ratio (%) | Days -5, 1, 3, 5, 6, 8, 10 & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via bio-electrical impedance analysis.
Changes in body composition: Body Mass (kg) | Days -5, 1, 6, & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via DXA.
Changes in body composition: Fat Mass (kg) | Days -5, 1, 6, & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via DXA.
Changes in body composition: Percent Body Fat (%) | Days -5, 1, 6, & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via DXA.
Changes in body composition: Bone Mineral Content (g) | Days -5, 1, 6, & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via DXA.
Changes in body composition: Bone Mineral Density (g/cm^2) | Days -5, 1, 6, & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via DXA.
Changes in body composition: Fat Free Mass (kg) | Days -5, 1, 6, & 11
  Assessment of alterations in body mass and body composition following short-term energy balance and energy deficit. Assessed via DXA.
Changes in Resting Metabolic Rate (kcal/day) | Days -5, 1, & 11.
  Assessment of alterations in resting metabolic rate following short-term energy balance and energy deficit.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Areta, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Areta JL, Burke LM, Camera DM, West DW, Crawshay S, Moore DR, Stellingwerff T, Phillips SM, Hawley JA, Coffey VG. Reduced resting skeletal muscle protein synthesis is rescued by resistance exercise and protein ingestion following short-term energy deficit. Am J Physiol Endocrinol Metab. 2014 Apr 15;306(8):E989-97. doi: 10.1152/ajpendo.00590.2013. Epub 2014 Mar 4. PMID 24595305
- [Background] Areta JL, Hopkins WG. Skeletal Muscle Glycogen Content at Rest and During Endurance Exercise in Humans: A Meta-Analysis. Sports Med. 2018 Sep;48(9):2091-2102. doi: 10.1007/s40279-018-0941-1. PMID 29923148
- [Background] Areta JL, Iraki J, Owens DJ, Joanisse S, Philp A, Morton JP, Hallen J. Achieving energy balance with a high-fat meal does not enhance skeletal muscle adaptation and impairs glycaemic response in a sleep-low training model. Exp Physiol. 2020 Oct;105(10):1778-1791. doi: 10.1113/EP088795. Epub 2020 Sep 7. PMID 32820838
- [Background] Civitarese AE, Carling S, Heilbronn LK, Hulver MH, Ukropcova B, Deutsch WA, Smith SR, Ravussin E; CALERIE Pennington Team. Calorie restriction increases muscle mitochondrial biogenesis in healthy humans. PLoS Med. 2007 Mar;4(3):e76. doi: 10.1371/journal.pmed.0040076. PMID 17341128
- [Background] Hall KD. Body fat and fat-free mass inter-relationships: Forbes's theory revisited. Br J Nutr. 2007 Jun;97(6):1059-63. doi: 10.1017/S0007114507691946. Epub 2007 Mar 19. PMID 17367567
- [Background] Hall KD, Chow CC. Estimating changes in free-living energy intake and its confidence interval. Am J Clin Nutr. 2011 Jul;94(1):66-74. doi: 10.3945/ajcn.111.014399. Epub 2011 May 11. PMID 21562087
- [Background] Hammond KM, Sale C, Fraser W, Tang J, Shepherd SO, Strauss JA, Close GL, Cocks M, Louis J, Pugh J, Stewart C, Sharples AP, Morton JP. Post-exercise carbohydrate and energy availability induce independent effects on skeletal muscle cell signalling and bone turnover: implications for training adaptation. J Physiol. 2019 Sep;597(18):4779-4796. doi: 10.1113/JP278209. Epub 2019 Aug 21. PMID 31364768
- [Background] Hawley JA, Morton JP. Ramping up the signal: promoting endurance training adaptation in skeletal muscle by nutritional manipulation. Clin Exp Pharmacol Physiol. 2014 Aug;41(8):608-13. doi: 10.1111/1440-1681.12246. PMID 25142094
- [Background] Holwerda AM, Bouwman FG, Nabben M, Wang P, van Kranenburg J, Gijsen AP, Burniston JG, Mariman ECM, van Loon LJC. Endurance-Type Exercise Increases Bulk and Individual Mitochondrial Protein Synthesis Rates in Rats. Int J Sport Nutr Exerc Metab. 2020 Mar 1;30(2):153-164. doi: 10.1123/ijsnem.2019-0281. Epub 2020 Feb 7. PMID 32035417
- [Background] Impey SG, Hearris MA, Hammond KM, Bartlett JD, Louis J, Close GL, Morton JP. Fuel for the Work Required: A Theoretical Framework for Carbohydrate Periodization and the Glycogen Threshold Hypothesis. Sports Med. 2018 May;48(5):1031-1048. doi: 10.1007/s40279-018-0867-7. PMID 29453741
- [Background] Rabol R, Svendsen PF, Skovbro M, Boushel R, Haugaard SB, Schjerling P, Schrauwen P, Hesselink MK, Nilas L, Madsbad S, Dela F. Reduced skeletal muscle mitochondrial respiration and improved glucose metabolism in nondiabetic obese women during a very low calorie dietary intervention leading to rapid weight loss. Metabolism. 2009 Aug;58(8):1145-52. doi: 10.1016/j.metabol.2009.03.014. Epub 2009 Jun 18. PMID 19454354
- [Background] Rhoads TW, Clark JP, Gustafson GE, Miller KN, Conklin MW, DeMuth TM, Berres ME, Eliceiri KW, Vaughan LK, Lary CW, Beasley TM, Colman RJ, Anderson RM. Molecular and Functional Networks Linked to Sarcopenia Prevention by Caloric Restriction in Rhesus Monkeys. Cell Syst. 2020 Feb 26;10(2):156-168.e5. doi: 10.1016/j.cels.2019.12.002. Epub 2020 Jan 22. PMID 31982367
- [Background] Smiles WJ, Areta JL, Coffey VG, Phillips SM, Moore DR, Stellingwerff T, Burke LM, Hawley JA, Camera DM. Modulation of autophagy signaling with resistance exercise and protein ingestion following short-term energy deficit. Am J Physiol Regul Integr Comp Physiol. 2015 Sep;309(5):R603-12. doi: 10.1152/ajpregu.00413.2014. Epub 2015 Jul 1. PMID 26136534
- [Background] Whytock KL, Parry SA, Turner MC, Woods RM, James LJ, Ferguson RA, Stahlman M, Boren J, Strauss JA, Cocks M, Wagenmakers AJM, Hulston CJ, Shepherd SO. A 7-day high-fat, high-calorie diet induces fibre-specific increases in intramuscular triglyceride and perilipin protein expression in human skeletal muscle. J Physiol. 2020 Mar;598(6):1151-1167. doi: 10.1113/JP279129. Epub 2020 Feb 14. PMID 31958145